CLINICAL TRIAL: NCT04083183
Title: Targeted Astatine-211-Labeled BC8-B10 Monoclonal Antibody as Reduced Intensity Conditioning for Nonmalignant Diseases
Brief Title: Total Body Irradiation and Astatine-211-Labeled BC8-B10 Monoclonal Antibody for the Treatment of Nonmalignant Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1005632; NCI-2019-05727 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9524 (Other: Fred Hutch / University of Washington Cancer Consortium); P01HL122173-01 (NIH)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-Malignant Neoplasm
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Whole-Body Irradiation; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (astatine 211,fludarabine,cyclophosphamide,TBI,HCT) (Experimental): Patients receive astatine At 211 anti-CD45 monoclonal antibody BC8-B10 IV on any day between days -10 and -7, fludarabine IV on days -6 to -2, cyclophosphamide IV over 1 hour on days -6 to -5 and 3 to 4, and thymoglobulin IV over 4-6 hours on days -4 to -2. Patients undergo TBI on day -1 and hematopoietic cell transplant on day 0. Beginning day 5, patients also receive mycophenolate mofetil PO or IV thrice daily every 8 hours up to day 35 if no GVHD present and sirolimus PO daily until day 365. Patients undergo blood sample collection and may undergo bone marrow aspiration throughout the study.
  Interventions: Biological: Astatine At 211 Anti-CD45 Monoclonal Antibody BC8-B10; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Lapine T-Lymphocyte Immune Globulin; Radiation: Total-Body Irradiation; Procedure: Hematopoietic Cell Transplantation; Drug: Mycophenolate Mofetil; Drug: Sirolimus; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Astatine At 211 Anti-CD45 Monoclonal Antibody BC8-B10 — Given IV
  Other Names: Astatine 211-Labeled Anti-CD45 Monoclonal Antibody BC8-B10; Astatine At 211 MAb BC8-B10; At 211 Anti-CD45 Monoclonal Antibody BC8-B10; At 211 MAb BC8-B10; APAMISTAMAB-B10-ASTATINE AT-211
Drug: Fludarabine — Given IV
  Other Names: 2-Fluorovidarabine; 21679-14-1; 9-Beta-D-arabinofuranosyl-2-fluoro-9H-purin-6-amine; 9-Beta-D-arabinofuranosyl-2-fluoroadenine; Fluradosa; 2-Fluoro-9-beta-arabinofuranosyladenine; 2-Fluorovidarabine, 21679-14-1
Drug: Cyclophosphamide — Given IV
  Other Names: Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclostin; Cyclostine; Cytoxan; WR-138719
Biological: Lapine T-Lymphocyte Immune Globulin — Given IV
  Other Names: Anti-thymocyte Globulin Rabbit; Grafalon; Rabbit Anti-Human Thymocyte Globulin (RATG); Rabbit Anti-Thymocyte Globulin; Rabbit Antithymocyte Globulin; Rabbit ATG; rATG; Thymoglobulin
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; TOTAL BODY IRRADIATION; Whole Body Irradiation; Whole-Body Irradiation; SCT_TBI
Procedure: Hematopoietic Cell Transplantation — Undergo hematopoietic cell transplantation
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF; 115007-34-6
Drug: Sirolimus — Given PO
  Other Names: RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This phase I/II trial studies the best dose of total body irradiation with astatine-211 BC8-B10 monoclonal antibody for the treatment of patients with nonmalignant diseases undergoing hematopoietic cell transplant. Radiation therapy uses high energy gamma rays to kill cancer cells and shrink tumors. Astatine-211-labeled BC8-B10 monoclonal antibody is a monoclonal antibody, called anti-CD45 monoclonal antibody BC8-B10, linked to a radioactive/toxic agent called astatine 211. Anti-CD45 monoclonal antibody BC8-B10 is attached to CD45 antigen positive cancer cells in a targeted way and delivers astatine 211 to kill them. Giving astatine-211 BC8-B10 monoclonal antibody and total-body irradiation before a donor stem cell transplant may help stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive astatine At 211 anti-CD45 monoclonal antibody BC8-B10 intravenously (IV) on any day between days -10 and -7, fludarabine IV on days -6 to -2, cyclophosphamide IV over 1 hour on days -6 to -5 and 3 to 4, and thymoglobulin IV over 4-6 hours on days -4 to -2. Patients undergo TBI on day -1 and hematopoietic cell transplant on day 0. Beginning day 5, patients also receive mycophenolate mofetil orally (PO) or IV thrice daily every 8 hours up to day 35 if no GVHD present and sirolimus PO daily until day 365. Patients undergo blood sample collection and may undergo bone marrow aspiration throughout the study.

After completion of study treatment, patients are followed up at 1 and 2 years and then periodically for up to 5 years.

Note: National Heart, Lung, and Blood Institute (NHLBI) funding for this study ended in 2022.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and < 50 years
* Nonmalignant disease treatable by allogeneic hematopoietic cell transplantation (HCT). Patients with a nonmalignant disease that is not clearly defined must be approved by the principal investigator (PI)
* Karnofsky score >= 70
* Patients must have normal elastography
* If ferritin is elevated, patient must have less than 7 mg/g liver iron concentration on liver T2 magnetic resonance imaging (MRI)
* Patients should have an official gastrointestinal (GI) consult prior to the transplant for full evaluation
* DONOR INCLUSION
* HLA matched related donor that is genotypically or phenotypically identical for HLA-A, -B, -C, -DRB1, -DQB1. Phenotypic identity must be confirmed by high-resolution typing. Sibling donors are preferred over other relationships
* Unrelated donor.

  * Matched for HLA-A, -B, -C, -DRB1, and DQB1 by high-resolution typing; OR
  * Mismatched for a single HLA-class 1 allele or HLA-DQB1 antigen or allele by high-resolution typing.

Note: A donor homozygous for one allele only at HLA-A, B, C, DRB1, or DQB1 is allowed (1 antigen mismatch for graft versus host disease [GVHD], 0 antigen mismatch for graft-rejection). In the case of a recipient who is homozygous at one locus, the mismatch is not allowed to be at that locus (0 antigen mismatch for GVHD, 1 antigen mismatch for graft-rejection)

* HLA haploidentical donor. There must be one shared HLA-haplotype based on inheritance. The noninherited haplotype is allowed to be mismatched at any or all of these loci: HLA-A, B, C, DRB1 or DQB1.
* Donor selection guideline recommendations: in the case where there are multiple donor options, donors should be selected based on the following priority numbered below:

  * Related donor genotypically HLA-matched
  * Related donor phenotypically HLA-matched
  * Unrelated donor HLA-matched
  * Unrelated donor with single allele level mismatch at class 1 (HLA-A, -B, or -C). For example, HLA-A02:01 versus HLA-A 02:02
  * Unrelated donor with single allele level mismatch at DQB1
  * HLA-haploidentical donor Note: We require that the donor testing be performed by a United States Clinical Laboratory Improvement Amendment (CLIA) approved laboratory. In the very rare case where the donor testing is not able to be performed in a CLIA approved laboratory, or there is confirmatory testing that needs to be performed, or for any donor identified from Europe and at risk for Creutzfeldt-Jakob Disease (CJD), we note this on the donor screening form and require that the unrelated donor medical director or the attending physician approves the use of the donor HPC-A product under urgent medical need

Exclusion Criteria:

* Patients with Fanconi Anemia
* Impaired cardiac function as evidenced by ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%) or cardiac insufficiency requiring treatment or symptomatic coronary artery disease. Patients with a shortening fraction of < 26% may be enrolled if approved by a cardiologist. In addition, patients with poorly controlled hypertension on multiple anti-hypertensive medications, symptomatic coronary artery disease, or patients on cardiac medications for antiarrhythmic or inotropic effects are excluded
* Impaired pulmonary function as evidenced by carbon monoxide diffusing capability test (DLCO) < 35% of predicted or receiving supplemental continuous oxygen. In addition, if patients are unable to perform pulmonary function tests, then O2 saturation < 92% on room air
* Impaired renal function as evidenced by estimated creatinine clearance less than 50 ml/min or serum creatinine > 2 x upper normal limit or dialysis-dependent. Serum creatinine value must be within 28 days prior to start of conditioning

  * The creatinine clearance may be estimated by the Cockcroft-Gault formula
* Impaired liver function as evidenced by abnormal hepatic function within 2 months prior to the astatine-211 infusion date defined as a total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) > 2 times the upper limit of normal (with the exception of elevated total bilirubin level, predominantly indirect bilirubin, in patients with hemoglobinopathy due to acute and/or chronic hemolysis). In addition, patients with the following liver abnormalities are excluded: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease
* An uncontrolled infection requiring deferral of conditioning as recommended by an infectious disease specialist. A viral upper respiratory tract infection does not constitute an uncontrolled infection in this context
* Patients who are known to be positive for HIV (human immunodeficiency virus)
* Women of childbearing potential who are pregnant or breast-feeding
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Allergy to murine-based monoclonal antibodies
* Known contraindication to radiotherapy
* DONOR EXCLUSION
* Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before hematopoietic cell transplantation (HCT). If the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive. For those patients with an HLA class I allele or class II allele or antigen mismatch or haploidentical donors, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results. A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2028-01-09 (Estimated); Study Completion 2028-01-09 (Estimated)

PRIMARY OUTCOMES:
Graft rejection (arm A) | Up to 5 years post-transplant
  Defined as establishment of < 5% donor chimerism of CD3+ T cells and <5% donor chimerism of CD33+ myeloid cells at day 80-100 after hematopoietic cell transplant (HCT) following an human leukocyte antigen (HLA)-matched related or unrelated graft or an unrelated graft with a single HLA-class 1 allele mismatch or DQB1 antigen or allele mismatch.
Graft rejection (arm B) | Up to 5 years post-transplant
  Defined as establishment of < 5% donor chimerism of CD3+ T cells and < 5% donor chimerism of CD33+ myeloid cells at day 80-100 after HCT following an HLA-haploidentical related donor or an unrelated donor mismatched for a single HLA-class 1 antigen or a single HLA-DRB1 allele.

SECONDARY OUTCOMES:
Transplant related mortality | At day 100 post-transplant
Overall survival | At 1 year post-transplant
Rate of acute graft versus host disease (GVHD) | At day 100 post-transplant
Rate of chronic GVHD | At 1 year post-transplant
Donor chimerism | At day 28, day 84, and 1 year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Vo, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No